CLINICAL TRIAL: NCT03062956
Title: Randomized, Placebo-Controlled Study of Safety, Tolerability, Preliminary Pharmacokinetics and Pharmacodynamics of Single Ascending Oral Doses of MYK-491 in Healthy Adult Volunteers
Brief Title: A Single Ascending Dose Study Assessing the Safety, Tolerability, PK and PD of MYK-491
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MyoKardia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MYK-491-001
Record Dates: First submitted 2017-02-16; First posted 2017-02-24 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized 6:2 to MYK-491:placebo within each cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single oral dose of MYK-491 (Experimental): single-dose, oral suspension
  Interventions: Drug: MYK-491 or placebo
- Single oral dose of placebo (Placebo Comparator): single-dose, oral suspension
  Interventions: Drug: MYK-491 or placebo

INTERVENTIONS:
Drug: MYK-491 or placebo — Oral suspension

SUMMARY:
Up to 72 healthy volunteers will be given a single dose of MYK-491 or placebo and be monitored for safety and tolerability over a 7 day period.

DETAILED DESCRIPTION:
Up to 72 healthy volunteers will be given a single dose of MYK-491 or placebo and be monitored for safety and tolerability over a 7 day period. After the 28 day screening period, the eligible subject will be admitted to the clinical site and will receive a single dose of study drug or placebo. Subjects will be confined to the clinical site for five days (Day -1 to Day 4) and will return to the clinic on Day 7 for a safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Weight between 60 and 90 kg inclusive
* Resting heart rate of < 80 beats per minute
* Documented LVEF greater than or equal to 55% during Screening
* Normal electrocardiogram (ECG) at Screening
* Normal acoustic windows on transthoracic echocardiograms at Screening
* All safety laboratory parameters within normal limits at Screening
* History or evidence of another clinically significant disorder, in the opinion of the investigator.

Exclusion Criteria:

* Active infection
* History of coronary artery disease
* History of malignancy with the exception of in situ cervical cancer more than 5 years prior to Screening or surgically-excised non-melanomatous skin cancers more than 2 years prior to Screening
* Positive serology tests at screening
* Current use of tobacco or nicotine-containing products exceeding 10 per day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessments will include treatment emergent AEs and SAEs, ECG recordings, vital signs, hs-troponin 1 concentrations, laboratory abnormalities and physical exam abnormalities | 7 days

SECONDARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) | 7 days
Maximum observed plasma concentration (Tmax) | 7 days
Area under the plasma concentration-time curve (AUC) | 7 days
First-order terminal elimination half-life (t1/2) | 7 days
Mean retention time (MRT) | 7 days

OTHER OUTCOMES:
The change from baseline in LVFS, LVEF, LVSV and SET by TTE | 7 days
SET while using photoplethysmography | 7 days
Relationship between MYK-491 plasma concentrations/PK parameters and PD parameters | 7 days
Plasma concentrations of metabolites of MYK-491 in plasma and urine | 7 days
Relationship between MYK-491 plasma concentration and QTc interval | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MD, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No